CLINICAL TRIAL: NCT06019559
Title: A Randomized, Placebo-Controlled, Double-Blind 13-Week Study to Evaluate the Safety, Tolerability, and Weight Loss Efficacy of K-757 Alone and in Combination With K-833 in Participants Who Are Obese
Brief Title: A Study to Evaluate the Safety, Tolerability, and Weight Loss Efficacy of K-757 Alone and in Combination With K-833
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kallyope Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-757 P006
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- K-757+K-833 (Experimental)
  Interventions: Drug: K-757 120 mg BID and K-833 100 mg BID
- K-757 alone (Experimental)
  Interventions: Drug: K-757 120 mg BID and matching placebo to K-833
- Placebo to K-757 and K-833 (Experimental)
  Interventions: Drug: Matching placebo to K-757 and matching placebo to K-833

INTERVENTIONS:
Drug: K-757 120 mg BID and K-833 100 mg BID — K-757 was titrated to the maintenance dose of 120 mg twice daily (BID) by Day 22. K-833 was initiated at 100 mg once daily in the morning (QAM) and was titrated to the maintenance dose of 100 mg BID on Day 8.
  Both administered orally.
  Arms: K-757+K-833
Drug: K-757 120 mg BID and matching placebo to K-833 — K-757 was titrated to the maintenance dose of 120 mg twice daily (BID) by Day 22.
  Both administered orally.
  Arms: K-757 alone
Drug: Matching placebo to K-757 and matching placebo to K-833 — Both administered orally.
  Arms: Placebo to K-757 and K-833

SUMMARY:
This is a study to evaluate the safety and efficacy of K-757 alone and in combination with K-833 versus placebo in participants who are obese.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the trial procedures and agree to participate by providing written informed consent prior to trial related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
2. Be willing and able to comply with the study schedule of visits, all trial procedures and restrictions, including following study diet requirements.
3. Be a male or female, age 18 to 70 years, inclusive, at the time of signing informed consent.
4. Have a body mass index (BMI) of 30.0 to <40.0. kg/m2, inclusive.
5. History of at least one self-reported unsuccessful dietary effort to lose body weight.
6. Be weight stable (<5% variation) over the last 3 months (by subject report).
7. Be a nonsmoker or has smoked ≤10 cigarettes per week for at least 3 months and agrees not to exceed this for the duration of study participation; has not used other nicotine containing products (e.g. other forms of tobacco, nicotine patch, e cigarettes, vapes) for at least 3 months and agrees to abstain from such products throughout study participation.
8. Meet the following requirements:

   1. Is a male who agrees to all of the following:

      * To use an appropriate method of contraception, including a condom which must include spermicidal cream or jelly, from the first dose of study drug until 14 days after the last dose of study drug. A male subject who had a vasectomy procedure must follow the same restrictions as a non vasectomized man.
      * If partner is pregnant, to use a condom
      * To not donate sperm from the first dose of study drug until 14 days after the last dose of study drug.

      OR
   2. Is a female who is of non-childbearing potential defined by at least 1 of the following criteria:

      * Postmenopausal (aged >45 years and with a minimum of 12 months of spontaneous amenorrhea with a Screening serum follicle-stimulating hormone (FSH) level in the menopausal range established for the central laboratory.
      * Post hysterectomy, bilateral oophorectomy or bilateral salpingectomy, based on the subject's recall of their medical history.

      OR
   3. Is a female of reproductive potential and:

      * agrees to not donate eggs from the first dose of study drug until 14 days after the last dose of study drug.
      * agrees to remain abstinent from heterosexual activity or
      * agrees to use (or have their partner use) a birth control method that is highly effective and has low user dependency from the first dose of study drug until 14 days after the last dose of study drug. Acceptable methods of birth control are:

        * Progestogen-only implant (e.g. etonogestrel implant)
        * Intrauterine device (IUD)
        * Intrauterine hormone-releasing system (IUS)
        * Bilateral tubal occlusion
        * Vasectomized partner

Exclusion Criteria:

Glycemia related:

1. Has a hemoglobin A1c (HbA1c) ≥6.5% (48 mmol/mol) as measured by the central laboratory at screening.
2. Has a history of clinically significant endocrine disease including T2DM. Note: A history of hypothyroidism does not require exclusion if the subject has been on a stable dose of thyroid hormone replacement (thyroxine) for at least 3 months prior to screening and the screening thyroid-stimulating hormone (TSH) is within the central laboratory normal range.
3. Has a history of type 1 or type 2 diabetes mellitus.
4. Had treatment with any glucose-lowering agent(s) within 90 days before screening.

   Obesity related:
5. Had treatment with any medication approved for the treatment of obesity or any investigational agent being tested for obesity treatment within the past 6 months before screening.
6. Has been treated with/used any other medication, supplement, or device for the purpose of promoting weight loss (regardless of whether they are approved or promoted for the purpose of weight loss) in the 90 days prior to screening.
7. Treatment with any glucagon-like peptide-1 (GLP-1) receptor agonist in the prior 6 months.
8. Participation in an organized weight reduction program (e.g. Weight Watchers) within 90 days of screening.
9. Had a previous or has a planned (during the trial period) obesity treatment with surgery or a weight loss device. Note: Prior liposuction and/or abdominoplasty are not exclusionary if performed >2 years before screening).
10. Has uncontrolled thyroid disease, defined as thyroid stimulating hormone (TSH) outside (above or below) the reference range of the central laboratory at screening or has any history of Grave's disease.
11. Obesity is induced by an endocrine disorder (e.g. Cushing's disease).

    Mental health:
12. Has a history of major depressive disorder within 2 years before screening unless all of the following criteria are met:

    1. the depressive disorder has always been unipolar (no history of mania or hypomania)
    2. in the opinion of the investigator, depressive symptoms have been stable and well controlled for ≥ 2 years prior to screening.
    3. any anti-depressant drug-treatment regimens (medications and doses) have been stable for ≥6 months prior to screening.
13. Has any history of other severe psychiatric disorder (e.g., schizophrenia, bipolar disorder) that was not clearly attributable to an intercurrent event/life circumstance, self-limited and fully resolved ≥1 year prior to screening.
14. On the screening Patient Health Questionnaire-9 (PHQ-9), has an overall score ≥15 or has a score >0 for Question # 9 (Thoughts that you would be better off dead or of hurting yourself).
15. Has any lifetime history of suicide attempt or suicidal behavior. Note: Suicidal behavior includes any acts/preparation toward making a suicide attempt whether the attempt is never initiated or is initiated but interrupted by self or another person.
16. Use of any anti-psychotic agents for any purpose within 2 years before screening.
17. Use of prohibited classes of anti-depressant agents, for any purpose, within 6 months of screening. Note: Use of allowable classes of anti-depressant agents is permitted only if the anti-depressant regimen (agents and doses) has been stable for ≥6 months prior to screening and is not anticipated to change during the trial period.

    General Safety:
18. Has a recent history (within the past 3 years of the screening visit) or current diagnosis of clinically significant hematological, immunological, renal, respiratory, neurologic, or genitourinary abnormalities or diseases.
19. Has a recent history (within past 3 years of the screening visit) or current diagnosis of any of the following GI (gastro intestinal) related diseases: intestinal obstruction, GI perforation, adhesions, Clostridium difficile colitis or have had recent unexplained GI bleeding within 3 months prior to screening.
20. Has any history of pancreatitis (acute or chronic), gastroparesis, ischemic colitis, inflammatory bowel disease (IBD), or celiac disease.
21. Has any personal or first-degree relative history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
22. Has a screening estimated Glomerular Filtration Rate (eGFR) estimated with the Modification of Diet in Renal Disease (MDRD) equation of <60 ml/min/1.73 m2.
23. Has a history of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed if they have received treatment and follow-up consistent with local standard of care.
24. Has any history of cardiovascular disease including stable and unstable angina pectoris, myocardial infarction, transient ischemic attack, stroke, cardiac decompensation, clinically significant arrhythmias, clinically significant conduction disorders, or any history or heart failure.
25. Has any surgery scheduled for the duration of the trial, except for minor surgical procedures, in the opinion of the investigator.
26. Has a history of human immunodeficiency virus (HIV) infection.
27. Has any active liver disease other than non-alcoholic fatty liver disease (NAFLD), or any gallbladder disease that has been active/symptomatic within 6 months of screening.
28. Has a positive test result for hepatitis B surface antigen (Ag), hepatitis C virus antibody, or HIV antibody, at the Screening Visit. Note: Participants with positive hepatitis B virus or hepatitis C virus serology may be enrolled if quantitative polymerase chain reaction for hepatitis B virus or hepatitis C virus ribonucleic acid is negative.
29. Has alanine aminotransferase or aspartate aminotransferase (ALT or AST) of >2.0X upper limit of normal (ULN) or total bilirubin >1.5X ULN at the Screening visit. Note: An isolated bilirubin >1.5X ULN is acceptable if bilirubin is fractionated, and direct bilirubin is within the laboratory normal range.
30. Has serum amylase or lipase >1.2X the ULN at the Screening visit.
31. Has a triglycerides value of >600mg/dL at the Screening visit (if value is ≥600 mg/dL and the sample was obtained in the non-fasted state, a repeat fasting determination may be obtained to assess eligibility).
32. Has a corrected QT interval to Fridericia's formula (QTcF) >450 milliseconds (msec) for males and >470 msec for females at screening.
33. Has a mean value for triplicate semi-recumbent systolic blood pressure >160 mmHg and/or diastolic blood pressure (BP) >95 mmHg measured after at least 10 minutes at rest at the Screening Visit.

    Note: If a subject's BP is exclusionary on the first triplicate assessment at the Screening visit, they may have 1 repeat triplicate BP assessment at that visit after another rest of at least 10 minutes.

    If a participant's BP is exclusionary on 2 assessments at the Screening visit, the investigator can, at their discretion, adjust and/or add anti-hypertensive medications and re-assess triplicate BP up to twice prior to dosing at the Randomization visit (Visit 2). Anti-hypertensive regimens must be ≤2 agents that do not include verapamil.

    If a participant's BP is exclusionary at the Screening visit and the Randomization visit (Visit 2), they must be excluded.
34. Has known history or suspected abuse of alcohol or recreational drugs at Screening.
35. Has excessive consumption of alcohol within 6 months prior to screening (>14 drinks/week for men and >7 drinks/week for women, where l drink= 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) or use of soft drugs (such as marijuana or any substances containing tetrahydrocannabinol (THC) or cannabidiol (CBD)) within 3 months prior to Screening, or hard drugs (such as cocaine) within 6 months prior to Screening.
36. Has a positive drug screen at Screening.
37. Has known or suspected hypersensitivity to trial product(s) or related products.
38. Has a history of multiple significant and/or any severe allergies (e.g., food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
39. Has previous participation in this trial. Participation is defined as signed informed consent.
40. Has participated in any clinical trial of an approved or non-approved investigational medicinal product within 90 days before screening.
41. Had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the Screening Visit.
42. Is a female who is pregnant, breast-feeding or intends to become pregnant during the planned course of the study. Note: Participants must have a negative serum pregnancy test (β-human chorionic gonadotropin (β-hCG)) performed by the central laboratory prior to enrollment in the study and prior to the randomization visit.
43. Is currently in violation of study requirements for prohibited and permissible concomitant medications or is anticipated to violate these requirements during study participation.
44. Has any disorder, unwillingness or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol.
45. Is unable or unwilling to follow the study nutritional and physical activity counseling and to refrain from alternative lifestyle modification strategies throughout study participation.
46. Is an employee or immediate family member (e.g., spouse, parent, child, sibling) of the Sponsor or study site.

Note: Rescreening/retesting is not permitted unless specified above.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Quest Research Institute, Farmington Hills, Michigan
  - ActivMed Practices and Research, LLC, Portsmouth, New Hampshire
  - Rochester Clinical Research, Rochester, New York
  - Medication Management, LLC (PharmQuest), Greensboro, North Carolina
  - Wilmington Health (Accellacare of Wilmington), Wilmington, North Carolina
  - Family Practice Center of Wadsworth, Inc dba New Venture Medical Research, Wadsworth, Ohio
  - AMR Norman, Norman, Oklahoma
  - Summit Headlands LLC, Portland, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Reading Hospital Clinical Trials Office, West Reading, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Headlands Research - Brownsville, Brownsville, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Washington Center for Weight Management and Research, Inc., Arlington, Virginia
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- K-757 Alone: K-757 120 mg BID and matching placebo to K-833. Both Administered orally.
- K-757+K-833: K-757 120 mg BID and K-833 100 mg BID. Both administered orally.
Period: Overall Study
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
Started | 52 | 51 | 52
Completed | 43 | 45 | 44
Not Completed | 9 | 6 | 8
Not completed — Withdrawal by Subject | 7 | 6 | 5
Not completed — Lost to Follow-up | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized all modified intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833 | Total
Number analyzed (Participants) | 52 | 51 | 52 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 36 | 48 | 133
  >=65 years | 3 | 15 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.93) | 50.6 (14.84) | 49.0 (11.90) | 48.9 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 35 | 105
  Male | 17 | 16 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 10 | 28
  Not Hispanic or Latino | 44 | 40 | 42 | 126
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 11 | 22
  White | 45 | 44 | 41 | 130
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 51 | 52 | 155
Weight [Mean (Standard Deviation); unit: kg] | 100.21 (14.426) | 99.36 (13.979) | 100.03 (13.830) | 99.87 (13.994)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Body Weight (%) After 13 Weeks of Treatment
Time Frame: 13 weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: % Change from Baseline
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
Number analyzed (Participants) | 52 | 51 | 52
% Change from Baseline | -0.15 (0.562) | -1.57 (0.566) | -2.94 (0.587)
Statistical Analysis 1: Comparison: Placebo to K-757 and K-833 vs K-757 Alone; Test type: Superiority; p = 0.0756, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; MMRM model with gender, treatment, visit and treatment-by-visit interaction as fixed effect, and baseline body weight as a covariate
Statistical Analysis 2: Comparison: Placebo to K-757 and K-833 vs K-757+K-833; For the primary endpoint of percentage change from baseline in body weight, a sample size of 150 participants (stratified by gender and randomized 1:1:1 into three treatment arms) provided >95% power to detect a treatment difference of 4% weight reduction after 13 weeks of treatment with a 2-sided alpha of 0.05, assuming a standard deviation of 4% and 20% drop out; Test type: Superiority; p = 0.0008, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; (MMRM) model with gender, treatment, visit and treatment-by-visit interaction as fixed effect, and baseline body weight as a covariate

2. Secondary Outcome: The Proportion of Participants Achieving ≥5% Weight Loss After 13 Weeks of Treatment
Time Frame: 13 weeks
Population: Modified Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
Number analyzed (Participants) | 52 | 51 | 52
Participants | 6 | 9 | 11
Statistical Analysis 1: Comparison: Placebo to K-757 and K-833 vs K-757 Alone; Test type: Superiority; p = 0.8366, Regression, Logistic — The threshold for significance was p = 0.05
Statistical Analysis 2: Comparison: Placebo to K-757 and K-833 vs K-757+K-833; Test type: Superiority; p = 0.1848, Regression, Logistic — The threshold for significance was p = 0.05

3. Secondary Outcome: Absolute Change From Baseline in Body Weight (kg) After 13 Weeks of Treatment
Time Frame: 13 weeks
Population: Modified Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
Number analyzed (Participants) | 52 | 51 | 52
kg | -0.09 (0.582) | -1.64 (0.587) | -3.11 (0.609)
Statistical Analysis 1: Comparison: Placebo to K-757 and K-833 vs K-757 Alone; Test type: Superiority; p = 0.0616, Mixed Models Analysis — The threshold for significance was p = 0.05
Statistical Analysis 2: Comparison: Placebo to K-757 and K-833 vs K-757+K-833; Test type: Superiority; p = 0.0004, Mixed Models Analysis — The threshold for significance was p = 0.05

4. Secondary Outcome: Proportion of Participants Who Experienced 1 or More Treatment-emergent AEs
Description: This outcome is descriptive and no formal statistical analysis was performed.
Time Frame: 15 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
Number analyzed (Participants) | 52 | 51 | 52
Participants | 31 | 41 | 42

5. Secondary Outcome: Proportion of Participants Who Discontinued Study Medication Due to an AE
Description: This outcome is descriptive and no formal statistical analysis was performed.
Time Frame: 13 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
Number analyzed (Participants) | 52 | 51 | 52
Participants | 2 | 9 | 14

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Placebo to K-757 and K-833 | K-757 Alone | K-757+K-833
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 31/52 | 41/51 | 42/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo to K-757 and K-833 (N=52) | K-757 Alone (N=51) | K-757+K-833 (N=52)
Nausea (Gastrointestinal disorders) | 9 (9) | 15 (15) | 27 (27)
Constipation (Gastrointestinal disorders) | 2 (2) | 13 (13) | 19 (19)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (7) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 9 (9) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 4 (4)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 5 (5)
Fatigue (General disorders) | 2 (2) | 5 (5) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT06019559/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT06019559/SAP_001.pdf